CLINICAL TRIAL: NCT06676865
Title: Preoperative Prediction of Difficult Laryngoscopy in Diabetic Patients: Importance of the Palm Print Test
Status: Completed | Type: Observational
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Clinical Professor, Mongi Slim Hospital
Other Study IDs: Palm print test
Record Dates: First submitted 2024-10-22; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Difficult Laryngoscopy; Diabetes; Preoperative Period
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult Diabetic patients scheduled for surgery under general anesthesia.: Were included patients with known cases of diabetes mellitus, aged more than 18 years, undergoing surgery under general anesthesia with endotracheal intubation.
  This study excluded patients with physical or intellectual disabilities preventing cooperation, Malformations, trauma, tumors, or infections of the maxillofacial region and upper airways, a history of burns or cervicofacial irradiation, and neurosurgical conditions causing temporomandibular pseudoankylosis. Additional exclusions included patients with conditions causing hand joint stiffness (e.g., carpal tunnel syndrome, Dupuytren's disease, scleroderma, rheumatoid arthritis), restricted cervical mobility (due to osteoarthritis, ankylosing spondylitis, or cervical trauma), a history of difficult intubation as well as pregnancy (including up to six weeks postpartum)
  Interventions: Diagnostic Test: the palm print test

INTERVENTIONS:
Diagnostic Test: the palm print test — The patient's dominant hand was pressed firmly against a blue ink pad, then onto a white sheet of paper without applying body weight. The palm prints were scored as follows:
  * Grade 0: All phalangeal areas visible
  * Grade 1: Deficiency in the interphalangeal areas of the 4th and 5th digits
  * Grade 2: Deficiency in the interphalangeal areas of the 2nd to 5th digits
  * Grade 3: Only the tips of the digits visible The palm print test was scored from 0 to 3. Grades 2 and 3 were considered indicators of difficult intubation.

SUMMARY:
The investigators assessed upper airway management at the pre-anaesthetic consultation using the usual clinical criteria. On the day before surgery, diabetic patients were assessed for the palm print sign to predict difficult laryngoscopy. After induction of anesthesia, laryngoscopy was performed with a Macintosh metal laryngoscope blade. At this stage of the study, patients were categorized into two groups: difficult and easy laryngoscopy.

DETAILED DESCRIPTION:
During pre-anesthesia consultation, all participants were assessed for airway conditions using usual clinical tests (Mallampati classification, Thyromental distance, mouth-opening test, upper lip biting test (ULBT), Head extension and Prayer sign). Demographic characteristics, diabetes duration, Blood glucose regulation and diabetes-related complications were also recorded.

On the day before surgery, patients were assessed for the palm print sign during preoperative evaluation rounds. On the day of surgery, after an intravenous line (IV) and complete monitoring, induction of anesthesia was initiated, and a muscle relaxant was used to facilitate intubation. Laryngoscopy was performed with a Macintosh metal laryngoscope blade by an anesthesiologist who had more than 2 years of intubation experience. McGrath® videolaryngoscope, McCoy laryngoscope, LMA Fastrack®, or i-gel® airway were kept ready for emergency situations. At this stage of the study, patients were categorized into two groups: difficult and easy laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus
* aged more than 18 years
* undergoing surgery under general anesthesia with endotracheal intubation.

Exclusion Criteria:

* physical or intellectual disabilities preventing cooperation
* Malformations, trauma, tumors, or infections of the maxillofacial region and upper airways,
* a history of burns or cervicofacial irradiation
* neurosurgical conditions causing temporomandibular pseudoankylosis.
* hand joint stiffness (e.g., carpal tunnel syndrome, Dupuytren's disease, scleroderma, rheumatoid arthritis)
* restricted cervical mobility (due to osteoarthritis, ankylosing spondylitis, or cervical trauma),
* a history of difficult intubation
* pregnancy (including up to six weeks postpartum)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Were included adult patients with diabetes mellitus undergoing surgery under general anesthésia with intubation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Difficult laryngoscopy | after induction of anesthesia and during laryngoscopy
  Cormack and Lehane graded I to IV. Grades III or IV showed difficult laryngoscopy.

SECONDARY OUTCOMES:
Difficult intubation | at induction of anesthesia
  Need of more than 2 laryngoscopies to intubate the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi Slim University Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No